CLINICAL TRIAL: NCT04448821
Title: A Clinical Trial to Evaluate the Effect of Nilotinib on the Pharmacokinetics and Pharmacodynamics of Metformin in Healthy Male Adults
Brief Title: A Clinical Trial to Evaluate the Effect of Nilotinib on the PK/PD of Meformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyewon Chung (Other)
Responsible Party: Sponsor-Investigator, Hyewon Chung, Clinical Assistant Professor, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NM-DDI
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: metformin; Period 2: metformin + nilotinib
  Interventions: Drug: Metformin; Drug: Metformin + Nilotinib
- Sequence B (Experimental): Period 1: metformin + nilotinib; Period 2: metformin
  Interventions: Drug: Metformin; Drug: Metformin + Nilotinib

INTERVENTIONS:
Drug: Metformin — Single administration of metformin
Drug: Metformin + Nilotinib — Coadministration of metformin and nilotinib

SUMMARY:
The aim of the study is to evaluate the effect of nilotinib on the pharmacokinetics and pharmacodynamics of metformin in healthy male adults

DETAILED DESCRIPTION:
Pharmacokinetics and pharmacodynamics of metformin without coadministration of nilotinib will be compared with those after administration of nilotinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 50 years
* Subjects with body mass index (BMI) between 18.5 and 29.9 kg/m2 and weight more than 50 kg
* Subjects who agree with performing contraception during the study
* Subjects who provides written informed consent

Exclusion Criteria:

* Subjects who have a current or prior history of cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, skin, psychiatric, or neurological diseases that is clinically significant
* Subjects who have clinically significant allergic history or allergy to metformin, nilotinib, or other components of drug
* Subjects with history of galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption
* Subjects with hypokalemia or hypomagnesemia at screening
* Subjects with QTcF > 450 or clinically significant findings on 12-lead ECG at screening
* Subjects with fasting plasma glucose lower than 70 mg/dL or upper than 126 mg/dL at screening
* Subjects who have history of gastrointestinal surgery
* Subjects with creatinine clearance ≤ 60mL/min at screening
* Subjects with AST or ALT ≥ 2-folds of upper normal limit
* Subjects who reports less than 12 points on taste test at screening
* Subjects who have administrated drugs that are known to cause significant drug-drug interaction with investigational drugs within 2 weeks prior to dosing
* Whole blood donation within 60 days prior to dosing, or apheresis donation within 20 days prior to dosing, or received blood donation within 30 days prior to dosing
* Subjects who participated in a previous clinical trial within 6 months prior to dosing
* Subjects with a history of alcohol abuse
* Subjects who are determined as unsuitable for clinical trial participation by investigator's decision

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours post-dose
  maximum concentration
AUCinf | 24 hours post-dose
  Area under the concentration-time curve from time of administration extrapolated to infinity
Gmax | 3 hours from 2 hour post-dose
  maximum glucose level during oral glucose tolerance test
AUGC | 3 hours from 2 hour post-dose
  Area under the concentration-time curve during oral glucose tolerance test

SECONDARY OUTCOMES:
Taste test | 7 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Chung, MD, PhD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

REFERENCES:
- [Background] Graham GG, Punt J, Arora M, Day RO, Doogue MP, Duong JK, Furlong TJ, Greenfield JR, Greenup LC, Kirkpatrick CM, Ray JE, Timmins P, Williams KM. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 2011 Feb;50(2):81-98. doi: 10.2165/11534750-000000000-00000. PMID 21241070
- [Background] Chen EC, Liang X, Yee SW, Geier EG, Stocker SL, Chen L, Giacomini KM. Targeted disruption of organic cation transporter 3 attenuates the pharmacologic response to metformin. Mol Pharmacol. 2015 Jul;88(1):75-83. doi: 10.1124/mol.114.096776. Epub 2015 Apr 28. PMID 25920679
- [Background] Kwon EY, Chung JY, Park HJ, Kim BM, Kim M, Choi JH. OCT3 promoter haplotype is associated with metformin pharmacokinetics in Koreans. Sci Rep. 2018 Nov 16;8(1):16965. doi: 10.1038/s41598-018-35322-6. PMID 30446679
- [Background] Lapczuk-Romanska J, Busch D, Gieruszczak E, Drozdzik A, Piotrowska K, Kowalczyk R, Oswald S, Drozdzik M. Membrane Transporters in Human Parotid Gland-Targeted Proteomics Approach. Int J Mol Sci. 2019 Sep 28;20(19):4825. doi: 10.3390/ijms20194825. PMID 31569384
- [Background] Lee N, Duan H, Hebert MF, Liang CJ, Rice KM, Wang J. Taste of a pill: organic cation transporter-3 (OCT3) mediates metformin accumulation and secretion in salivary glands. J Biol Chem. 2014 Sep 26;289(39):27055-27064. doi: 10.1074/jbc.M114.570564. Epub 2014 Aug 8. PMID 25107910
- [Background] Minematsu T, Giacomini KM. Interactions of tyrosine kinase inhibitors with organic cation transporters and multidrug and toxic compound extrusion proteins. Mol Cancer Ther. 2011 Mar;10(3):531-9. doi: 10.1158/1535-7163.MCT-10-0731. Epub 2011 Jan 20. PMID 21252289
- [Background] Rhee SJ, Choi Y, Lee S, Oh J, Kim SJ, Yoon SH, Cho JY, Yu KS. Pharmacokinetic and pharmacodynamic interactions between metformin and a novel dipeptidyl peptidase-4 inhibitor, evogliptin, in healthy subjects. Drug Des Devel Ther. 2016 Aug 10;10:2525-34. doi: 10.2147/DDDT.S110712. eCollection 2016. PMID 27570447
- [Background] Jang K, Chung H, Yoon JS, Moon SJ, Yoon SH, Yu KS, Kim K, Chung JY. Pharmacokinetics, Safety, and Tolerability of Metformin in Healthy Elderly Subjects. J Clin Pharmacol. 2016 Sep;56(9):1104-10. doi: 10.1002/jcph.699. Epub 2016 Feb 22. PMID 26710683
- [Background] Hwang CS, Kim JW, Al Sharhan SS, Kim JW, Cho HJ, Yoon JH, Kim CH. Development of a Gustatory Function Test for Clinical Application in Korean Subjects. Yonsei Med J. 2018 Mar;59(2):325-330. doi: 10.3349/ymj.2018.59.2.325. PMID 29436203